CLINICAL TRIAL: NCT03063944
Title: Phase I Trial of OPB-111077 in Combination With Decitabine and Venetoclax for the Treatment of AML Refractory to or Ineligible for Intensive Chemotherapy
Brief Title: STAT Inhibitor OPB-111077, Decitabine and Venetoclax in Treating Patients With Acute Myeloid Leukemia That Is Refractory, Relapsed or Newly Diagnosed and Ineligible for Intensive Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16C.773; JT 10092 (Other: JeffTrial Number)
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Injections; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (STAT inhibitor OPB-111077, venetoclax, decitabine) (Experimental): INDUCTION CYCLE 1: Patients receive STAT inhibitor OPB-111077 PO QD on days 1-28, and venetoclax PO QD on days 4-28 of cycle 1. Patients also receive decitabine IV over approximately 1 hour on days 4-8 of cycle 1. Patients who achieve complete remission (CR) after 1 cycle move on to Maintenance, and patients who do not achieve a CR move on to Cycle 2.
  INDUCTION CYCLE 2: Patients receive STAT inhibitor OPB-111077, venetoclax, and decitabine as in Induction Cycle 1. Patients who achieve CR, CRi, PR, or stable disease (or clinically significant hematologic improvement as determined by the investigator) move on to Maintenance.
  MAINTENANCE: Patients receive STAT inhibitor OPB-111077, venetoclax, and decitabine as in Induction Cycle 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: STAT Inhibitor OPB-111077; Drug: Decitabine; Drug: Venetoclax; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: STAT Inhibitor OPB-111077 — Given PO
  Other Names: OPB-111077
Drug: Decitabine — Given IV
  Other Names: 2'-Deoxy-5-azacytidine; 4-Amino-1-(2-deoxy-beta-D-erythro-pentofuranosyl)-1,3,5-triazin-2(1H)-one; 2353-33-5; 5-Aza-2'-deoxycytidine; 5-Aza-2'deoxycytidine; 5-Aza-2-deoxycytidine; 5-Azadeoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Drug: Venetoclax — Given PO
  Other Names: 1257044-40-8; 4-(4-((2-(4-Chlorophenyl)-4; 4-dimethylcyclohex-1-en-1-yl)methyl)piperazin-1-yl)-N-((3-nitro-4-((tetrahydro-2H-pyran-4-ylmethyl)amino)phenyl)sulfonyl)-2-(1H-pyrrolo(2,3-b)pyridin-5-yloxy)benzamide; ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of STAT inhibitor OPB-111077 when given together with decitabine and venetoclax in treating patients with acute myeloid leukemia that does not respond to treatment (refractory), has come back (relapsed), or is newly diagnosed and ineligible for intensive chemotherapy. STAT inhibitor OPB-111077 and decitabine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as venetoclax, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving STAT inhibitor OPB-111077, decitabine, and venetoclax may work better in treating patients with acute myeloid leukemia compared to decitabine alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability of STAT inhibitor OPB-111077 (OPB-111077) in combination with decitabine and venetoclax.

SECONDARY OBJECTIVES:

I. To describe any preliminary efficacy of OPB-111077 in combination with decitabine and venetoclax in patients with acute myeloid leukemia (AML).

II. To measure adenosine triphosphate (ATP) generation and perform metabolomics in patients with AML who are receiving OPB-111077, decitabine, and venetoclax.

III. To assess apoptosis and proliferation assays in patients with AML who are receiving OPB-111077, decitabine, and venetoclax.

OUTLINE: This is a dose escalation study of STAT inhibitor OPB-111077.

INDUCTION CYCLE 1: Patients receive STAT inhibitor OPB-111077 orally (PO) once daily (QD) on days 1-28, and venetoclax PO QD on days 4-28 of cycle 1. Patients also receive decitabine intravenously (IV) over approximately 1 hour on days 4-8 of cycle 1. Patients who achieve complete remission (CR) after 1 cycle move on to Maintenance, and patients who do not achieve a CR move on to Cycle 2.

INDUCTION CYCLE 2: Patients receive STAT inhibitor OPB-111077, venetoclax, and decitabine as in Induction Cycle 1. Patients who achieve CR, complete remission with incomplete hematologic recovery (CRi), partial remission (PR), or stable disease (or clinically significant hematologic improvement as determined by the investigator) move on to Maintenance.

MAINTENANCE: Patients receive STAT inhibitor OPB-111077, venetoclax, and decitabine as in Induction Cycle 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic evidence of high risk acute myeloid leukemia defined as one of the following:

  * Non-M3 AML refractory to standard primary induction therapy
  * Non-M3 AML relapsed after (i) any standard induction therapy (ii) any number of standard or experimental salvage therapies
  * Newly diagnosed non-M3 AML not eligible for intensive induction chemotherapy
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* Subjects must have a life expectancy of at least 4 weeks
* Subjects must be able to consume oral medication
* Subjects must have recovered from the toxic effects of any prior chemotherapy to= < grade 1 (except alopecia)
* Creatinine clearance (CrCL) >= 45
* Total bilirubin =< 2 x upper limit of normal (ULN)
* Serum glutamate pyruvate transaminase (SGPT) alanine aminotransferase (ALT) =< 2 x ULN
* Negative pregnancy test for women with child-bearing potential
* Patients must be able to sign consent and be willing and able to comply with scheduled visits, treatment plan and laboratory testing

Exclusion Criteria:

* Subjects with FAB M3 (t(15;17)(q22;q21)[PML-RARalpha]) are not eligible
* Subjects must not be receiving any chemotherapy agents (except hydroxyurea); intrathecal methotrexate and cytarabine are permissible
* Subjects must not be receiving growth factors, except for erythropoietin
* Subjects with a "currently active" second malignancy, other than non-melanoma skin cancer, carcinoma in situ of the cervix, resected incidental prostate cancer (staged pT2 with Gleason score =< 6 and postoperative prostate-specific antigen [PSA] < 0.5 ng/mL), or other adequately treated carcinoma-in-situ are ineligible; patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for >= 1 year
* Subjects with uncontrolled high blood pressure, unstable angina, symptomatic congestive heart failure (New York Heart Association [NYHA] class 3), myocardial infarction within the past 6 months or serious uncontrolled cardiac arrhythmia are not eligible
* Subjects with other severe concurrent disease which in the judgment of the investigator would make the patient inappropriate for entry into this study are ineligible
* Subjects must not have evidence of active leukemia in the central nervous system (CNS)
* Subjects must not have received any investigational agents within 14 days or 5 half-lives (whichever is longer) of study entry
* Subjects must not be pregnant or breastfeeding; pregnancy tests must be obtained for all females of child-bearing potential; pregnant or lactating patients are ineligible for this study; males or women of childbearing potential may not participate unless they have agreed to use an effective contraceptive method (defined as hormonal contraceptives, intrauterine devices, surgical contraceptives, or condoms)
* Subjects who have uncontrolled infection are not eligible; patients must have any active infections under control; fungal disease must be stable for at least 2 weeks before study entry
* Subjects with bacteremia must have documented negative blood cultures prior to study entry
* Subjects who are suitable for and willing to receive standard intensive induction therapy
* Subjects who are candidates for allogeneic transplantation, have a suitable donor, and are willing to undergo transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 4, non-hematologic dose limiting toxicities assessed by National Cancer Institute Common Toxicity Criteria for Adverse Events version 5.0 | Up to 2 years
  Data analysis will be descriptive. All estimates of dose-specific rates (e.g., response and toxicity) will be presented with corresponding confidence intervals using the exact method. The method of Atkinson and Brown will be used for any rate related to definition of dose limiting toxicity, due to two-stage sampling. The method of Conover will be used otherwise.

SECONDARY OUTCOMES:
Metabolomics as determined by bone marrow biopsy | At the end of Cycle 1 (each cycle is 28 days)
  Data analysis will be descriptive.
Adenosine triphosphate (ATP) generation as determined by bone marrow biopsy | At the end of Cycle 1 (each cycle is 28 days)
  Data analysis will be descriptive.
Apoptotic rate in blood and bone marrow assessed by apoptosis assays | At the end of Cycle 1 (each cycle is 28 days)
  Data analysis will be descriptive.
Cellular proliferation in blood and bone marrow assessed by proliferation assays | At the end of Cycle 1 (each cycle is 28 days)
  Data analysis will be descriptive.
Complete response as determined by bone marrow biopsy | At the end of Cycle 1 (each cycle is 28 days)
  Data analysis will be descriptive
Complete response in the absence of total platelet recovery determined by bone marrow biopsy | At the end of Cycle 1 (each cycle is 28 days)
  Data analysis will be descriptive

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Kasner, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/